CLINICAL TRIAL: NCT07004803
Title: The Effect of Virtual Reality on Pain and Fear Levels of Children With Primary Immunodeficiency Applying Intravenous Immunoglobulin During Intravenous Access: A Crossover Randomized Controlled Trial
Brief Title: Virtual Reality on Pain and Fear Levels of Children With Primary Immunodeficiency
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Hatice Dönmez (Other)
Collaborators: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Sponsor-Investigator, Dr. Hatice Dönmez, Assistant professor, Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: KMU-SBF-HD-01; 16-M-24 (Other Grant/Funding Number: Karamanoglu Mehmetbey Unversity)
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Primary Immunodeficiency Diseases (PID)
Keywords: Children; Virtual Reality; Primary Immunodeficiency; Nursing care; Administration, Intravenous
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental)
  Interventions: Other: Virtual reality video watching
- Tablet group (Active Comparator)
  Interventions: Other: Tablet video watching

INTERVENTIONS:
Other: Virtual reality video watching — The children in the VR experimental group of the study will be subjected to the clinic's routine venipuncture procedure and the video-watching intervention with virtual reality headset. Routine care includes informing the child and parents about the procedure and questions that strengthen communication and distract attention. For example, it consists of questions such as 'How old are you?', 'Do you go to school?', 'Can you tell me the name of your favorite friend?'. Virtual reality headset will be introduced to the child before the procedure and information about how to use them will be given. After the measurements, intravenous access will be started. During the procedure, children will be shown a roller coaster video on virtual reality headset. The video-viewing process will be started 2 minutes before the venipuncture procedure. The video viewing time is planned to last an average of 4 minutes. Measurements were made during and after the procedure
  Arms: Virtual reality group
Other: Tablet video watching — The children in the experimental group of the study will be subjected to the clinic's routine venipuncture procedure and the video-watching intervention with Tablet. Routine care includes informing the child and parents about the procedure and questions that strengthen communication and distract attention. For example, it consists of questions such as 'How old are you?', 'Do you go to school?', 'Can you tell me the name of your favorite friend?'. Tablet will be introduced to the child before the procedure and information about how to use them will be given. After the measurements, intravenous access will be started. During the procedure, children will be shown a roller coaster video on tablet. The video-viewing process will be started 2 minutes before the venipuncture procedure. The video viewing time is planned to last an average of 4 minutes. Measurements were made during and after the procedure.
  Arms: Tablet group

SUMMARY:
In this study, it is aimed to investigate the effect of virtual reality and tablet video viewing intervention on pain and fear levels and vital signs of children during peripheral venous catheter placement for intravenous immunoglobulin (IVIG) administration.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 4-11
* Being followed up with the diagnosis of Primary Immunodeficiency for at least 6 months
* To accept participation in the study voluntarily
* No additional chronic disease other than primary immunodeficiency

Exclusion Criteria:

* Organ failure is present
* Having a mental deficiency
* Having a disability to use VR Glasses
* Children with fever (|>37.5 C0)
* Children with severe dehydration

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Children's Fear Scale | 5 minutes
Wong-Baker Pain Scale | 5 minutes
Children's Emotional Manifestation Scale | 5 minutes

SECONDARY OUTCOMES:
Vital Signs | 5 minutes
  Pulse, oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No